CLINICAL TRIAL: NCT00811590
Title: Pilot Study of mTOR Inhibitor Therapy for Treatment of Intestinal Polyps in Peutz-Jeghers Syndrome
Brief Title: Pilot Study of mTOR Inhibitor Therapy in Peutz-Jeghers Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was ended early due to low enrollment.
Sponsor: University of Utah (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI26943
Record Dates: First submitted 2008-11-17; First posted 2008-12-19 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Peutz-Jeghers Syndrome
Keywords: Cancer; Polyps
MeSH Terms: conditions — Peutz-Jeghers Syndrome; Neoplasms; Polyps | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus is a novel derivative of rapamycin. Everolimus has been in clinical development since 1996 as an immunosuppressant in solid organ transplantation. Since 2003, RAD001 is approved in Europe (trade name: Certican) via the Mutual Recognition Procedure (MRP) for the prevention of organ rejection in patients with renal and cardiac transplantation. Certican is also approved in Australia, South Africa, the Middle East, Central and South America, the Caribbean and some Asian countries.
  Everolimus is being investigated as an anticancer agent based on its potential to act
  * directly on the tumor cells by inhibiting tumor cell growth and proliferation
  * indirectly by inhibiting angiogenesis leading to reduced tumor vascularity (via potent inhibition of tumor cell VEGF production and VEGF-induced proliferation of endothelial cells.
  Other Names: everolimus, Certican, Afinitor

SUMMARY:
Pilot study, Open-label, Phase II study of Everolimus.

Objective:

To determine if Everolimus can diminish large gastrointestinal polyps in patients with Peutz-Jeghers Syndrome.

Methodology:

Polyp size and number will be compared to baseline by FDG-PET and CT and 12 months after treatment with Everolimus. Since this is a pilot study, the polyps prior to treatment will serve as the controls.

DETAILED DESCRIPTION:
Peutz-Jeghers Syndrome is a hereditary polyposis condition in which hamartomatous tumors develop in many tissues of the body. These tumors are benign but frequently cause gastrointestinal obstruction and bleeding beginning in the 2nd-3rd decades of life necessitating surgical intervention. Unfortunately, a recent study showed that the lifetime risk of cancers that arise in Peutz-Jeghers Syndrome is 85% by age 70 years and is 60% by age 60 years (Hearle et al., 2006).

A working definition of PJS has been suggested by Giardiello et al ,1987(www.genetests.com):

* For individuals with a histopathologically confirmed hamartoma, a definite diagnosis of PJS requires two of the following three findings:

  * Family history consistent with autosomal dominant inheritance
  * Mucocutaneous hyperpigmentation (although this can fade with age)
  * Small-bowel polyposis
* For individuals without histopathologic verification of hamartomatous polyps, a probable diagnosis of PJS can be made based on the presence of two of the three clinical criteria above.
* For individuals without a family history of PJS, diagnosis depends upon the presence of two or more histologically verified Peutz-Jeghers-type hamartomatous polyps (Tomlinson & Houlston 1997).
* For individuals with a first-degree relative with PJS, presence of mucocutaneous hyperpigmentation is sufficient for presumptive diagnosis.

Recently, rapamycin (Rapamune, Wyeth), an FDA-approved drug for use in orthotopic transplant recipients, was successfully used in an off-label study of 5 individuals with a related condition called tuberous sclerosis in which the patients had subependymal giant cell astrocytomas that caused significant and insidious neurological problems such as hydrocephalus and seizures (Franz, et al. 2006). All astrocytoma lesions exhibited regression with treatment of oral rapamycin and in one case, necrosis. Treatment was well tolerated and may offer an alternative to operative therapy in tuberous sclerosis. Tuberous sclerosis is caused by germline mutations in the tuberous sclerosis 1 or 2 genes. These genes encode proteins that function downstream of STK11, the gene that is mutated in Peutz-Jeghers Syndrome. Mutations of STK11 or TSC1/2 leads to activation of mTOR (mammalian target of rapamycin). Dysregulation of mTOR has been demonstrated in several types of cancers and clinical trials are underway to see if inhibition of mTOR will be of benefit to a variety of cancer patients. A recent trial showed efficacy of everolimus in advanced renal cancer (Hudes, et al. 2007).

All of these studies will be performed on an outpatient basis.

ELIGIBILITY:
Inclusion Criteria:

Yes/No (Response of "no" = patient ineligible)

1. Patients who are 18 years or older with a clinical or genetic diagnosis of Peutz-Jeghers Syndrome.
2. Patient has one or more intestinal polyps ≥ 5mm in maximum diameter by contrast enhanced CT scan that is not clinically indicated for removal or is beyond the reach of a push endoscope.
3. Minimum of two weeks since any major surgery.
4. Patient has had colonoscopy within the past 24 months and did not have high-grade dysplasia or colorectal cancers.
5. WHO performance status £ 2
6. Adequate bone marrow function as shown by: ANC ≥ 1.5 x 109/L, Platelets ≥ 100 x 109/L, Hgb > 9 g/dL
7. Adequate liver function as shown by: serum bilirubin ≤ 1.5 x upper limit of normal (ULN), and serum transaminases activity ≤ 2.5 x ULN.
8. Patients must be able to provide written informed consent.

Exclusion Criteria:

Yes/No (Response of "yes" = patient ineligible)

1. Prior treatment with any investigational drug within the preceding 4 weeks
2. Chronic treatment with systemic steroids or another immunosuppressive agent
3. Patients should not receive immunization with attenuated live vaccines during study period or within one week of study entry
4. Uncontrolled brain or leptomeningeal metastases, including patients who continue to require glucocorticoids for brain or leptomeningeal metastases
5. Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin.
6. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

   1. Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction ≤ 6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia
   2. Severely impaired lung function
   3. Uncontrolled diabetes as defined by fasting serum glucose >1.5x ULN
   4. Any active (acute or chronic) or uncontrolled infection/ disorders.
   5. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy
   6. Liver disease such as cirrhosis, or severe hepatic impairment (Child-Pugh class C)
   7. A known history of HIV seropositivity
   8. Impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of everolimus (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection)
   9. Patients with an active, bleeding diathesis or on oral anti-vitamin K medication
7. Women who are pregnant or breast feeding, or women/men able to conceive and unwilling to practice an effective method of birth control throughout the trial and for 8 weeks after the last dose of study drug. (Women of childbearing potential must have a negative pregnancy test). Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
8. Male patients whose sexual partner(s) are WOCBP who are not willing to use adequate contraception during the study and for 9 weeks after the end of treatment.
9. Patients who have received treatment with an mTor inhibitor in the past 6 months.
10. Patients with a known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus) or to its excipients

Patients who can not undergo FDG-PET are eligible to participate in this study for the purpose of the primary endpoint. Patient with the following will be excluded from FDG-PET piece of the study.

1. Patients cannot have a serum glucose level greater than 200 mg/dl for FDG-PET imaging
2. Patients who are too claustrophobic to undergo FDG-PET imaging
3. Patients who will require conscious sedation to undergo FDG-PET imaging.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall W Burt, MD, Principal Investigator — Huntsman Cancer Institute; Scott Kuwada, MD, Study Chair — University of Hawaii
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Patients: All patients enrolled/eligible.
Period: Overall Study
Arm/Group | All Patients
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6667 (18.71719)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Size of Intestinal Polyps
Time Frame: 24 months
Population: Due to small enrollment number, analysis was not possible.
Groups:
- All Patients: All enrolled/eligible patients.
Arm/Group | All Patients
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Patients
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes